CLINICAL TRIAL: NCT05759208
Title: A Phase 2, Multi-center, Randomized, Double-Masked and Placebo-Controlled Study Evaluating the Efficacy and Safety of OK-101 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye Disease
Brief Title: The Study Evaluating the Efficacy and Safety of OK-101 in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Okyo Pharma Ltd (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-110-0018
Record Dates: First submitted 2023-02-23; First posted 2023-03-08 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double mask and placebo-controlled
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Experimental): OK-101 Placebo Ophthalmic Solution (vehicle): 1 drop BID in each eye (N = ~80)
  Interventions: Drug: Placebo
- Low Dose OK-101 (Experimental): 0.05% OK-101 Ophthalmic Solution: 1 drop BID in each eye (N = ~80)
  Interventions: Drug: OK-101
- High-Dose OK-101 (Experimental): 0.1% OK-101 Ophthalmic Solution: 1 drop BID in each eye (N = ~80)
  Interventions: Drug: OK-101

INTERVENTIONS:
Drug: OK-101 — Ophthalmic Solution
  Arms: High-Dose OK-101; Low Dose OK-101
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the safety and efficacy of OK-101 Ophthalmic Solution to placebo for the treatment of the signs and symptoms of dry eye.

DETAILED DESCRIPTION:
Subjects eligible to be randomized will receive either OK-101 or placebo to be administered bilaterally twice daily (BID) for 12 weeks (from Visit 2 to Visit 5). During a 14-day study run-in period (for the purpose of subject selection) prior to randomization, all subjects will receive Placebo Ophthalmic Solution (vehicle) bilaterally BID.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age;
2. Provide written informed consent;
3. Be willing and able to comply with all study procedures;
4. Have a patient-reported history of dry eye for at least 6 months prior to Visit 1;
5. Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1;
6. Have a best corrected visual acuity (BCVA) of 0.7 logarithm of the minimum angle of resolution (logMAR) or better (Snellen equivalent score of 20/100 or better) in each eye at Visit 1;
7. Report a score of ≥ 2 according to the Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire in at least one of the dry eye symptoms at Visits 1 and 2;
8. Have a Schirmer's Test score of ≤ 10 mm and ≥ 1 mm at Visits 1 and 2;
9. Have a corneal fluorescein staining score of ≥ 2 in at least one region according to the Ora Calibra® Corneal and Conjunctival Staining Scale for Grading of Fluorescein Staining in at least one region in one eye at Visits 1 and 2 and a central score ≥ 1 in the same eye;
10. Have a total lissamine green conjunctival score of ≥ 2, based on the sum of the temporal and nasal regions pre-CAE® at Visits 1 and 2;
11. Have a conjunctival redness score ≥ 1 according to the Ora Calibra® Conjunctival Redness for Dry Eye Scale in at least one eye at Visits 1 and 2 pre- CAE;
12. Demonstrate in the same eye(s) a response to the CAE at Visits 1 and 2 as defined by:

    1. Having at least a ≥1 point increase in fluorescein staining in the inferior region in at least one eye following CAE® exposure;
    2. Reporting an Ocular Discomfort score ≥3 at 2 or more consecutive time points in at least one eye during CAE® exposure (if a subject has an Ocular Discomfort rating of 3 at time = 0 for an eye, s/he must report an Ocular Discomfort rating of 4 for two consecutive measurements for that eye). Note: a subject cannot have an Ocular Discomfort score of 4 at time = 0);
13. Have at least one eye, the same eye, satisfy all criteria for 8, 9, 10, 11 and 12 above;
14. A negative urine pregnancy test if female of childbearing potential (those who are not surgically sterilized [bilateral tubal ligation, hysterectomy or bilateral oophorectomy] or post- menopausal [12 months after last menses]) and must use adequate birth control through the study period. For non-sexually active females, abstinence may be regarded as an adequate method of birth control.

Exclusion Criteria:

1. Have any clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction, ocular rosacea, lid margin inflammation, or active ocular allergies that require therapeutic treatment, or currently using tetracyclines (e.g., doxycycline, minocycline, tetracycline) and/or in the opinion of the investigator may interfere with study parameters;
2. Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
3. Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
4. Have previously had laser-assisted in situ keratomileusis (LASIK) surgery, Photorefractive keratectomy (PRK), or small incision lenticule extraction (SMILE) within the last 12 months;
5. Have used Restasis®, Xiidra®, Cequa®, Tyrvaya®, serum tears, generic cyclosporine A, and EYSUVIS® within 30 days of Visit 1;
6. Have had any ocular and/or lid surgeries in the past 6 months or have any planned ocular and/or lid surgeries over the study period;
7. Any use of Lipiflow, thermopulsation, Meibomian gland expression or intense pulsed light treatment within 6 months of visit 1
8. Be using or anticipate using temporary punctal plugs during the study that have not been stable within 30 days of Visit 1 or have permanent punctal plugs or had surgical punctal occlusion;
9. Be currently taking any topical ophthalmic prescription (including medications for glaucoma) or over-the-counter solutions, artificial tears, gels or scrubs, and cannot discontinue these medications for the duration of the trial (excluding medications allowed for the conduct of the study); the respective wash-out periods are required for the following medications:

   1. Antihistamines (including ocular): 72 hours prior to Visit 1
   2. Oral aspirin or aspirin-containing products allowed if dose has been stable over past 30 days prior to Visit 1 and no change in dose is anticipated during the study period
   3. Corticosteroids or mast cell stabilizers (including ocular): 14 days prior to Visit 1
   4. Any medication (oral or topical) known to cause ocular drying that has not been administered as a stable dose for at least 30 days prior to Visit 1 and during the study
   5. Neurostimulators: 30 days prior to Visit 1
   6. Current use or planned use of Prokera® during study conduct or within 30 days prior to Visit 1
   7. All other topical ophthalmic preparations (including artificial tear substitutes) other than the study drops: 72 hours prior to Visit 1
10. Have an uncontrolled systemic disease;
11. Be a woman who is pregnant, nursing, or planning a pregnancy;
12. Be unwilling to submit a urine pregnancy test at Visit 1 and Visit 6 (or early termination visit) if of childbearing potential. Non-childbearing potential is defined as a woman who is permanently sterilized (e.g., has had a hysterectomy or tubal ligation), or is postmenopausal (without menses for 12 consecutive months);
13. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; intrauterine device; or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use adequate birth control as defined above for the remainder of the study;
14. Have a known allergy and/or sensitivity to the test article or its components;
15. Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
16. Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Total Corneal Fluorescein Staining | 85 days
  Total corneal fluorescein staining score of the study eye using the Ora Calibra® scale, measured by mean change from baseline (Visit 2 pre-CAE®) to Day 85 (Visit 6). Each of the 5 areas will be scored on a scale of 0 to 4 for a total minimum score of 0 to total maximum score of 20, with 0 being best and 20 being worst.
Ocular Discomfort Score | 85 days
  Ocular discomfort score of both eyes using the Ora Calibra® scale, measured by mean change from baseline (Visit 2 pre-CAE®) to Day 85 (Visit 6). Each eye will be scored separately on a scale from 1 to 4, with 1 being best and 4 being worst.

SECONDARY OUTCOMES:
Fluorescein Staining by Region | 85 days
  Fluorescein staining by region: central, superior, inferior, temporal, nasal, corneal sum, conjunctival sum, and total staining of each eye using the Ora Calibra® scale. Each of the 5 areas will be scored on a scale of 0 to 4 for a total minimum score of 0 to total maximum score of 20, with 0 being best and 20 being worst
Lissamine Green Staining by Region | 85 days
  Lissamine green staining by region: central, superior, inferior, temporal, nasal, corneal sum, conjunctival sum, and total staining of each eye using the Ora Calibra® scale. Each of the 5 areas will be scored on a scale of 0 to 4 for a total minimum score of 0 to total maximum score of 20, with 0 being best and 20 being worst.
Conjunctival Redness | 85 days
  Conjunctival redness of each eye using the Ora Calibra® scale. Each eye will be graded on a scale of 0 to 4, with 0 being best and 4 being worst.
Schirmer's Test | 85 days
  Schirmer's Test of each eye

CONTACTS AND LOCATIONS:
Overall Officials: Raj Patil, PhD, Study Director — Okyo Pharma Ltd
Locations (6):
- United States (6):
  - Eye Research Foundation, Newport Beach, California
  - Vision Institute, Colorado Springs, Colorado
  - Butchertown clinical Trials, Louisville, Kentucky
  - Andover Eye Associates, Andover, Massachusetts
  - Core Inc., Shelby, North Carolina
  - Total Eye Care, PA, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No